CLINICAL TRIAL: NCT04001231
Title: A Phase 1, Open-Label Study to Evaluate Single and Multiple Dose Pharmacokinetics, Safety, and Tolerability of Exenatide Once-Weekly Suspension in Chinese Patients With Type 2 Diabetes Mellitus
Brief Title: Study of Exenatide Once-Weekly Suspension in Chinese Patients With Type 2 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study is stopped based upon strategic considerations impacting the clinical development of exenatide once-weekly suspension in China
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D5553C00008
Record Dates: First submitted 2019-05-07; First posted 2019-06-28 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes
Keywords: Pharmacokinetics; Safety; Tolerability; exenatide once weekly; Chinese
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Single group
Masking Description: Open-label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm of exenatide once-weekly suspension (Experimental): Exenatide once-weekly suspension via subcutaneous (SC) injection
  Interventions: Drug: Exenatide Once-Weekly Suspension

INTERVENTIONS:
Drug: Exenatide Once-Weekly Suspension — A single dose will be administered as 2.0-mg dose of exenatide onceweekly suspension via subcutaneous (SC) injection followed by blood samples be drawn for up to 168 hours after the first dose on Day 1 to assess single-dose PK for exenatide once-weekly suspension. Subsequently Patients will receive the second dose of the investigational product (IP) at Visit 6 (Day 8). Thereafter, patients will receive weekly (±1 day) doses of IP up to Visit 18 (Week 14).

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, tolerability, and safety of single and multiple doses of exenatide once-weekly suspension via subcutaneous (SC) injection using a pre-filled, single-dose autoinjector in male and female Chinese with type 2 diabetes.

DETAILED DESCRIPTION:
This is an open-label, single- and multiple-dose, PK study in Chinese subjects with type 2 diabetes mellitus. Up to 30 patients may initially be enrolled to target at least 20 patients completing the study. Up to 10 more patients (ie, 40 in total) may be subsequently recruited to replace patients who discontinue, provided such discontinuations are not due to significant (based on PI and Sponsor judgment) safety or tolerability issues. Eligible patients will receive their first 2.0-mg dose of exenatide once-weekly suspension via subcutaneous (SC) injection using a pre-filled, single-dose autoinjector at Visit 3 (Day 1).Blood samples will be drawn for up to 168 hours after the first dose on Day 1 to assess single-dose PK for exenatide once-weekly suspension. Patients will receive the second dose of the investigational product (IP) at Visit 6 (Day 8). Thereafter, patients will receive weekly (±1 day) doses of IP up to Visit 18 (Week 14). Intensive and extended PK sampling will be conducted after administration of the final dose (Dose 14) to assess multiple-dose PK for exenatide once-weekly suspension. Follow-up observations will be conducted at Visits 22 to 29 (Weeks 15 to 26), with the final follow-up at/after Visit 29 (Week 26 ±2 days). During follow-up period, Blood samples will be collected for PK analyses. Subjects will be monitored closely for adverse events throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study-specific procedures.
2. Male or female patients with T2DM treated with diet modification and exercise alone or in combination with a stable (in PI's opinion) regimen of metformin only for at least two months prior to screening. The T2DM diagnosis will be confirmed clinically by the PI, and should be consistent with the World Health Organization criteria for diagnosis and classification of diabetes
3. Between 20 to 75 years of age inclusive at Visit 1 (Screening)
4. The following criterion applies to females of child-bearing potential (not surgically sterilized and between menarche and 1-year postmenopause) only:

   1. Test negative for pregnancy at the time of screening.
   2. Intend not to become pregnant during the study.
   3. Are sexually inactive or have practiced a reliable method of birth control (for example, use of oral contraceptives or levonorgestrel, diaphragms with contraceptive jelly, cervical caps with contraceptive jelly, condoms with contraceptive foam, intrauterine devices, partner with vasectomy) for at least 6 weeks prior to screening.
   4. Agree to continue to use a reliable method of birth control (as determined by the PI) during the study and until 90 days after last dose.
5. Have a body weight of ≥45 kg and a body mass index (BMI) of 18.5 to 35 kg/m2 inclusive at Visit 1 (Screening).
6. Have clinical laboratory test results within the normal reference range for the population or study site, or with abnormalities deemed clinically insignificant by the PI. Abnormalities of plasma glucose (fasting ≤12.0 mmol/L and anytime≤15.0mmol/L), HbA1c (<10.5%), plasma lipids (TG<5.7 mmol/L), and urinary protein (with a range of trace < 2+ on dipstick) are acceptable.
7. Venous access sufficient to allow blood sampling as per the protocol.
8. Are reliable and willing to be available for the duration of the study and are willing to follow study procedures.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to bothAstraZeneca staff and/or staff at the study site, and direct family members).
2. Previous enrollment in the present study or have previously completed or withdrawn from any other study investigating exenatide.
3. Within 30 days of the initial dose of IP, have received treatment with a drug that has not received regulatory approval for any indication.
4. Known allergy or hypersensitivity to exenatide or any of the excipients contained in these agents (exenatide: sodium acetate buffer, mannitol, metacresol, MCT vehicle).
5. Previous treatment with exenatide or related GLP-1 receptor agonist compounds.
6. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, haematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
7. Systolic blood pressure (SBP) persistently (on ≥2 separate occasions) >160 mmHg on stable regimen of antihypertensive medication or >180 mmHg regardless of antihypertensive treatment.
8. History of, or currently have angina, revascularization, myocardial infarction, or heart failure.
9. Clinically significant peripheral vascular disease.
10. Evidence of poorly controlled T2DM or evidence of significant diabetes-related complications such as:

    1. Plasma glucose >12 mmol/L (fasting) or >15 mmol/L (anytime) at Visit 1 (Screening)
    2. HbA1c >10.5%
    3. History of hypoglycemic or hyperglycemic coma within 1 year prior to Visit 1 (Screening)
    4. History of active diabetic proliferative retinopathy or macular oedema
    5. Known significant autonomic neuropathy as evidenced by urinary retention, orthostatic hypotension, diabetic diarrhea, or gastroparesis
11. Two or more episodes of major hypoglycemia within 6 months prior to Visit 1 (Screening). See Section 5.2.8.1 for hypoglycemia classification.
12. Impaired renal function (serum creatinine >125 μ/mol/L in women, >132 μ/mol/L in men).
13. Liver disease, acute or chronic hepatitis, alanine aminotransferase (ALT/SGPT), or aspartate aminotransferase (AST) ≥3x upper limit of normal (ULN) of the reference range and total bilirubin level (TBL) ≥2xULN.
14. Evidence of hepatitis B and/or positive hepatitis B surface antigen.
15. Clinical symptoms associated with cholelithiasis (eg, cholecystitis or biliary colic), within 3 years of Visit 1 (Screening).
16. History of, or currently have acute or chronic pancreatitis, or have triglyceride concentrations ≥500 mg/dL at Visit 1 (Screening).
17. Have a serum calcitonin concentration ≥40 pg/mL at Visit 1 (Screening).
18. An abnormality in the 12-lead ECG that, in the opinion of the PI, increases the risks associated with participating in the study.
19. Evidence of significant active neuropsychiatric disease.
20. Evidence of current use of drugs of abuse or history of use within the past year.
21. Women who are lactating and/or breastfeeding.
22. Use of over-the-counter or prescription medication (other than thyroid replacement therapy, metformin, antihypertensive medication, lipid-lowering agents, aspirin, or paracetamol/acetaminophen) 7 and 14 days, respectively prior to dosing. If this situation arises, inclusion of an otherwise suitable patient may occur if permitted by the PI and Sponsor.
23. Significant active hematological disease and/or blood donation of more than 400 mL within the last 6 months.
24. An average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or patients unwilling to adhere to study alcohol restrictions (1 unit=360 mL of beer; 150 mL of wine; 45 mL of distilled spirits).
25. A personal or family history of medullary thyroid cancer or multiple endocrine neoplasia 2A or 2B.
26. Currently enrolled in any other clinical study.
27. Determined by the PI to be unsuitable for inclusion in this study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2021-07-02 (Estimated); Study Completion 2021-07-02 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations versus time profile of exenatide | Blood sample will be collected on Visit 3-6 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 7-17 (pre-dose). Visit 18-22 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 23-29 (once/visit).
  To evaluate the PK of single and multiple doses of exenatide once-weekly suspension in native Chinese patients with T2DM
Cmax | Blood sample will be collected on Visit 3-6 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 7-17 (pre-dose). Visit 18-22 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 23-29 (once/visit).
  Maximum plasma concentration directly from the observed concentration versus time data
tmax | Blood sample will be collected on Visit 3-6 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 7-17 (pre-dose). Visit 18-22 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 23-29 (once/visit).
  Time of maximum plasma concentration
AUC(0-8h) | Blood sample will be collected on Visit 3-6 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 7-17 (pre-dose). Visit 18-22 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 23-29 (once/visit).
  Area under the plasma concentration-time curve from zero (pre-dose) to time 8 h calculated by linear up/log down trapezoidal rule (following the first dose on Day 1)
AUC(0-168h) | Blood sample will be collected on Visit 3-6 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 7-17 (pre-dose). Visit 18-22 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 23-29 (once/visit).
  Area under the plasma concentration-time curve from zero (pre-dose) to time 168 h calculated by linear up/log down trapezoidal rule (following the first dose on Day 1)
AUCτ,ss | Blood sample will be collected on Visit 3-6 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 7-17 (pre-dose). Visit 18-22 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 23-29 (once/visit).
  Area under the plasma concentration-time curve over a dosing interval at steady state calculated by linear up/log down trapezoidal rule (following administration at Week 14)
Cav,ss | Blood sample will be collected on Visit 3-6 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 7-17 (pre-dose). Visit 18-22 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 23-29 (once/visit).
  Average plasma concentration at steady state calculated as AUCτ ,ss/τ (following administration at Week 14)
λ z | Blood sample will be collected on Visit 3-6 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 7-17 (pre-dose). Visit 18-22 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 23-29 (once/visit).
  Apparent terminal elimination rate constant (1/h) determined by linear regression of the terminal points of the log-linear concentration-time curve. Visual assessment will be used to identify the terminal linear phase of the concentration-time profile. A minimum of 3 data points and an Rsq of at least 0.800 will be used for determination. (following administration at Week 14)
t½ | Blood sample will be collected on Visit 3-6 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 7-17 (pre-dose). Visit 18-22 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 23-29 (once/visit).
  Apparent terminal half-life (h) determined as ln 2/λ z (following administration at Week 14)
CL/F | Blood sample will be collected on Visit 3-6 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 7-17 (pre-dose). Visit 18-22 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 23-29 (once/visit).
  Apparent total body clearance (L/h) calculated as dose/AUCτ,ss (following administration at Week 14)
Vss/F | Blood sample will be collected on Visit 3-6 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 7-17 (pre-dose). Visit 18-22 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 23-29 (once/visit).
  Apparent volume of distribution at steady state (following administration at Week 14)
Rac | Blood sample will be collected on Visit 3-6 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 7-17 (pre-dose). Visit 18-22 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 23-29 (once/visit).
  Accumulation ratio calculated as AUCτ,ss/AUC0-168h
Ctrough | Blood sample will be collected on Visit 3-6 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 7-17 (pre-dose). Visit 18-22 (pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 24, 72, 120, 168 hours post-dose). Visit 23-29 (once/visit).
  Trough plasma concentrations through the treatment period will be evaluated graphically to assess steady-state attainment

SECONDARY OUTCOMES:
Electrocardiograms (ECGs) | ECGs will be performed at Visit 1 (screening), Visit 3 (Day 1, pre-dose and 2 hours post-dose), Visit 18 (Week 14, Day 1, pre-dose and 2 hours post-dose) and Visit 29 (Week 26, follow-up)
  Safety as determined by analysis of 12-lead ECG. Routine 12-lead ECG will be done during study including test of heart rate, rhythm, P wave, QRS, PR interval, ST-T, QT interval.
Blood pressure (BP) | Blood pressure will be collected at Visit 1, Visit 3 (pre-dose, 2- and 24-hours post-dose), Visit 4 (post-dose), Visit 5 (post-dose), Visit 6-17 (pre-dose), Visit 18 (pre-dose, 2- and 24-hours post-dose), Visit 19-21 (post-dose), Visit 22-29
  Safety as determined by evaluation of supine blood pressure (systolic and diastolic) in mmHg.
Pulse rate | Pulse rate will be collected at Visit 1, Visit 3 (pre-dose, 2- and 24-hours post-dose), Visit 4 (post-dose), Visit 5 (post-dose), Visit 6-17 (pre-dose), Visit 18 (pre-dose, 2- and 24-hours post-dose), Visit 19-21 (post-dose), Visit 22-29
  Safety as determined by evaluation of supine pulse rate in beats per minute.
Body temperature | Body temperature will be collected at Visit 1, Visit 3 (pre-dose, 2- and 24-hours post-dose), Visit 4 (post-dose), Visit 5 (post-dose), Visit 6-17 (pre-dose), Visit 18 (pre-dose, 2- and 24-hours post-dose), Visit 19-21 (post-dose), Visit 22-29
  Safety as determined by evaluation of body temperature in Celsius degrees.
Safety and tolerability as determined by abnormality in clinical chemistry compared to baseline. | Blood sample will be collected at Visit 1 (screening), Visit 2 (admission, day -1), Visit 6 (Week2, pre-dose), Visit 8 (Week4, pre-dose), Visit 17 (Week13, pre-dose), Visit 23 (Week16, follow-up), Visit 29 (Week26, follow-up)
  Measurement of kidney function (e.g.urea, creatinine, Uric acid), liver function (ALP, ALT, AST, albumin, total bilirubin, direct bilirubin), lipid profile (total cholesterol, triglycerides, LDL, HDL), potassium and etc.
Safety and tolerability as determined by abnormality in hematology compared to baseline. | Blood sample will be collected at Visit 1 (screening), Visit 2 (admission, day -1), Visit 6 (Week2, pre-dose), Visit 8 (Week4, pre-dose), Visit 17 (Week13, pre-dose), Visit 23 (Week16, follow-up), Visit 29 (Week26, follow-up)
  Measurement of red blood cell count, white blood cell count, haemoglobin and platelets
Safety and tolerability as determined by abnormality in urinalysis compared to baseline. | Blood sample will be collected at Visit 1 (screening), Visit 2 (admission, day -1), Visit 6 (Week2, pre-dose), Visit 8 (Week4, pre-dose), Visit 17 (Week13, pre-dose), Visit 23 (Week16, follow-up), Visit 29 (Week26, follow-up)
  Measurement of leukocyte, red blood cells, protein and microscopy
Fasting blood glucose | Blood sample will be collected at Visit1, Visit3 (Day1, pre-dose), Visit4-5 (Day4, Day6, post-dose), Visit6-18 (Week2-14, pre-dose), Visit19 (Week14, Day4, post-dose) and Visit20 (Week14, Day6, post-dose), Visit22-26 (Week15-20) and Visit29 (Week26)
  Safety as determined by abnormality in blood glucose levels
Calcitonin | Blood sample will be collected at Visit1 (screening), Visit21 (Week14, Day7) and Visit29 (Week26, follow-up)
  Calcitonin levels will be measured per the study plan to determine the possible effect of exenatide once-weekly suspension on thyroid function.
Number of subjects with adverse events | Adverse event will be collected from Visit 1 (screening) to Visit 29 (Week 26, follow-up).
  Following categories will be collected and analyzed: any adverse event (AE), any AE causally related to investigational product (IP), serious adverse events (SAEs), SAEs causally related to IP, AEs with outcome of death, AEs leading to discontinuation of IP, and other significant AEs.
The presence and titer of anti-exenatide antibodies | Visit 3, Visit 6~18, Visit 21 and Visit 29 (once every visit)
  Historically, the small subset of exenatide concentrations associated with antibody titers >625 have been excluded from PK analyses due to evidence that these exenatide concentration measurements were unduly affected by negative interference from these antibodies in the exenatide bioanalytical method. Therefore the exenatide concentrations associated with antibody titers >625 may be excluded from the PK analysis.

OTHER OUTCOMES:
HbA1c | Blood sample will be collected at Visit1 (screening), Visit3 (Day1, pre-dose), Visit7 (Week 3, pre-dose), V10 (Week6, pre-dose), Visit13 (Week9, pre-dose), Visit16 (Week12, pre-dose), Visit21 (Week14, Day7, post-dose) and Visit29 (Week 26, follow-up)
  Exploratory evaluation of HbA1c after 2.0 mg exenatide given once weekly as a suspension in native Chinese patients with T2DM following single and multiple weekly SC injections

CONTACTS AND LOCATIONS:
Overall Officials: Quanying Zhang, Principal Investigator — Second Affiliated Hospital of Suzhou University

IPD SHARING:
Plan to Share IPD: Undecided